CLINICAL TRIAL: NCT00529737
Title: The Effect on Clip Markers Migration After Vacuum-Assisted Biopsy by Postprocedure Mammogram
Brief Title: Effect on Clip Markers After Vacuum-Assisted Biopsy by Postprocedure Mammogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0434
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Marker Clip Migration; Vacuum-Assisted Biopsy; Postprocedure Mammogram; Breast Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Post Procedure Mammogram Projection View A -- (view same projection as used in the biopsy procedure), then View B (view orthogonal projection to the first view).
  Interventions: Procedure: Breast Biopsy; Procedure: Post Procedure Mammogram
- Group 2 (Experimental): Post Procedure Mammogram Projection View B than View A
  Interventions: Procedure: Breast Biopsy; Procedure: Post Procedure Mammogram

INTERVENTIONS:
Procedure: Breast Biopsy — Stereotactic-guided breast biopsy via standard practice of care
Procedure: Post Procedure Mammogram — View of post-procedure mammogram same projection as used in the biopsy procedure (View A), and mammographic view orthogonal projection to the first view (View B).

SUMMARY:
Primary Objective:

- To perform a prospective study to determine if there is a different in the marker clip migration if the first post-biopsy mammogram was performed in the same projection as the core biopsy versus in the orthogonal projection.

DETAILED DESCRIPTION:
You are scheduled to have a biopsy because a lesion was seen on your mammogram. Sometimes, the lesion is completely removed during the biopsy. Therefore, a clip is usually placed to mark the biopsy site. If some of the tissue in this area needs to be removed by a surgeon at a later date, the clip will mark the area for your surgeon to remove.

All participants in this study will already be scheduled for a stereotactic biopsy with clip placement followed by a mammogram, as a part of the standard of care. You will need to sign a separate consent document for these procedures.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Blood (about 1 teaspoon) will be drawn for routine tests. Women who are able to have children must have a negative blood (about 1 teaspoon) pregnancy test before they can take part in this study.

If you are eligible and you choose to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two study groups. There will be an equal chance of being assigned to either group.

If you are assigned to Group 1, your breast will be compressed the same way as the breast was compressed during the biopsy in the first mammogram picture. In the second picture, your breast will be compressed the opposite way (a 90-degree rotation) from the way the first picture was done.

If you are assigned to Group 2, your breast will be compressed in a 90-degree rotation from the way the breast was compressed during your biopsy in the first mammogram picture. In the second picture, your breast will be compressed the same way as during the biopsy.

A researcher will review the mammogram to measure and record the distance of the biopsy clip from the biopsied lesion.

If your biopsy is benign (non-cancerous), you will return to the clinic for a mammogram once a year, as is standard of care. Researchers would like to review the mammogram that is taken 1 year after the biopsy in order to check to see if the clip has moved or stayed in the same place.

This is an investigational study. The clip used in this study is FDA approved. Up to 60 patients will take part in the study. All will be enrolled at M.D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* All patients who present to M. D. Anderson for a stereotactic guided 9 gauge vacuum-assisted breast biopsy and undergo stereotactic biopsy with biopsy clip deployment would be considered for the study.

Exclusion Criteria:

* If patient refuses biopsy or the biopsy is cancelled they will not be eligible.
* No biopsy clip is seen on the immediate postprocedure mammogram and no additional clip will be deployed.
* Pregnant women are excluded from the study.
* Patients who have had a previous biopsy or surgery in the same (ipsilateral) breast are excluded from the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Distance Traveled by Breast Clip | Pre-biopsy and post-biopsy mammograms, and follow up 1 year post biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Huong T. Le-Petross, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org